CLINICAL TRIAL: NCT02030002
Title: Use of a "Flash-free" Adhesive Resin for Orthodontic Bracket Bonding: a Clinical Study of Bonding Time, Bond Survival, and Adhesive Remnant Cleanup
Brief Title: Evaluation of a "Flash-free" Adhesive Resin for Orthodontic Bracket Bonding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1/2013
Record Dates: First submitted 2013-12-03; First posted 2014-01-08 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: Split-mouth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- APC Flash-Free Adhesive Coated Appliance System (Experimental): APC Flash-Free Adhesive Coated Appliance System
  Interventions: Device: APC Flash-Free Adhesive Coated Appliance System
- APC II Adhesive Coated Appliance System (Active Comparator): APC II Adhesive Coated Appliance System
  Interventions: Device: APC II Adhesive Coated Appliance System

INTERVENTIONS:
Device: APC Flash-Free Adhesive Coated Appliance System — APC Flash-Free Adhesive Coated Appliance System
  Arms: APC Flash-Free Adhesive Coated Appliance System
Device: APC II Adhesive Coated Appliance System — APC II Adhesive Coated Appliance System
  Arms: APC II Adhesive Coated Appliance System

SUMMARY:
The purpose of this study is to compare bonding time, bond survival, amount of adhesive remaining on the tooth surface after bracket debonding, and time required for adhesive remnant cleanup between a new "flash-free" and a conventional adhesive resin for orthodontic bracket bonding.

DETAILED DESCRIPTION:
Patients presenting for comprehensive orthodontic treatment with fixed appliances at the University of Minnesota, who are willing to participate, will be included in the initial study. Selection criteria will include full permanent dentition through the first molars, teeth with sound, non-carious buccal enamel and no pretreatment with chemical agents such as hydrogen peroxide, and no previous orthodontic treatment with fixed appliances. The patients will have their maxillary incisors, canines, and premolars bonded with ceramic orthodontic brackets pre-coated with a "flash-free" adhesive resin (Clarity Advanced Brackets APC flash-free, 3M Unitek, Monrovia, CA, USA) on one side and a conventional adhesive resin (Clarity Advanced Brackets APC II, 3M Unitek) on the other side. The side allocation and order of bonding will be randomized for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Full permanent dentition including incisors, canines, premolars, and first molars
* Teeth with sound, non-carious buccal enamel and no pretreatment with chemical agents such as hydrogen peroxide
* No previous orthodontic treatment with fixed appliances

Exclusion Criteria:

* Mental/emotional/developmental disability
* Cleft lip and/or palate, craniofacial anomaly, or syndrome
* Obvious oral hygiene issues such as excessive plaque accumulation, gingivitis, and/or pre-existing white spot lesions
* Prosthodontic or restored substrate extending on the labial surface of maxillary teeth
* Known allergies to any acrylates contained in the study materials

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Gruenheid, DDS, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Grunheid T, Larson BE. Comparative assessment of bonding time and 1-year bracket survival using flash-free and conventional adhesives for orthodontic bracket bonding: A split-mouth randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2018 Nov;154(5):621-628. doi: 10.1016/j.ajodo.2018.05.012. PMID 30384932
- [Derived] Grunheid T, Larson BE. A comparative assessment of bracket survival and adhesive removal time using flash-free or conventional adhesive for orthodontic bracket bonding: A split-mouth randomized controlled clinical trial. Angle Orthod. 2019 Mar;89(2):299-305. doi: 10.2319/030918-195.1. Epub 2018 Sep 19. PMID 30230375

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: This is a single-arm, split-mouth study. Participants receive both treatments at the same time. Participants had APC Flash-Free Adhesive Appliance System on one side of their mouth and APCII Adhesive Appliance System on the other side. The side allocation was randomized as follows. A randomization scheme with equal distribution of the two side allocations was generated using the online randomization tool at http://www.graphpad.com/quickcalcs. Allocation concealment was achieved with sequentially numbered, opaque sealed envelopes (SNOSE) containing the side allocation of the adhesives, which were prepared before the trial. An independent third party was responsible for opening the next envelope in sequence and implementing the randomization process.
Period: Enrollment
Arm/Group | All Participants
Started | 49
Completed | 44
Not Completed | 5
Not completed — Participant had change in treatment plan and no longer met the inclusion criteria | 1
Not completed — Participants signed consent, but enrollment was completed before their treatment began. | 4
Period: APC Flash-Free Adhesive Coated Appliance
Arm/Group | All Participants
Started | 44
Completed | 44
Not Completed | 0
Period: APC II Adhesive Coated Appliance System
Arm/Group | All Participants
Started | 44
Completed | 44
Not Completed | 0
Period: Follow-up
Arm/Group | All Participants
Started | 44
Completed | 42
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: All participants who received the treatment are included. The 4 participants who signed a consent, but did not begin treatment are excluded.
Groups:
- All Participants: This is a single-arm study. Participants receive both treatments at the same time. All participants are counted as one group at baseline.
Arm/Group | All Participants
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 45
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Bonding Time
Description: The time taken to bond each tooth was timed to the nearest second using a digital stopwatch. Timing was started after enamel surface preparation and stopped before light curing. Outcome reported in seconds.
Time Frame: At appliance placement, 30 minutes
Population: All participants who received the treatment are included in this analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | APC Flash-Free Adhesive Coated Appliance System | APC II Adhesive Coated Appliance System
Number analyzed (Participants) | 45 | 45
seconds | 42.5 (5.9) | 67.7 (5.9)

2. Primary Outcome: Bond Survival
Description: Bond failure (yes or no) was recorded at standardized appointments at intervals of 4 weeks. Outcome is reported as the cumulative number of failed bracket bonds across all participants at 1 year post-treatment.
Time Frame: 1 year post treatment
Population: Of the 45 participants who completed treatment, 43 completed the follow-up period and are included in this analysis.
Measure: Number; unit: failed bracket bonds
Arm/Group | APC Flash-Free Adhesive Coated Appliance System | APC II Adhesive Coated Appliance System
Number analyzed (Participants) | 43 | 43
failed bracket bonds | 8 | 2

3. Primary Outcome: Amount of Adhesive Remaining on the Tooth Surface After Bracket Debonding
Description: In case of a bond failure, the adhesive remnant index (ARI) was scored. The ARI is a point-based system ranking: 0, no adhesive left on the tooth; 1, less than half of the adhesive left on the tooth; 2, more than half of the adhesive left on the tooth; and 3, all adhesive left on the tooth.
Time Frame: At completion of treatment, 10 minutes.
Population: Of the 45 participants who completed treatment, 43 completed the follow-up period. One additional participant is excluded from this analysis due to a change in treatment plan that made them eligible according to the inclusion/exclusion criteria.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APC Flash-Free Adhesive Coated Appliance System | APC II Adhesive Coated Appliance System
Number analyzed (Participants) | 42 | 42
score on a scale | 2.53 (.36) | 2.29 (.4)

4. Primary Outcome: Time Required for Adhesive Remnant Cleanup
Description: If adhesive remained after bracket de-bonding, then the time required to remove the remnant adhesive was measured using a digital stop-watch. Outcome is reported in seconds.
Time Frame: At completion of treatment, 30 minutes.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | APC Flash-Free Adhesive Coated Appliance System | APC II Adhesive Coated Appliance System
Number analyzed (Participants) | 42 | 42
seconds | 167.3 (63.5) | 215.1 (79.8)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- APC Flash-Free Adhesive Coated Appliance System: APC Flash-Free Adhesive Coated Appliance System
  APC Flash-Free Adhesive Coated Appliance System: APC Flash-Free Adhesive Coated Appliance System
  Only the 45 participants who received treatment are included in the adverse event reporting.
- APC II Adhesive Coated Appliance System: APC II Adhesive Coated Appliance System
  APC II Adhesive Coated Appliance System: APC II Adhesive Coated Appliance System
  Only the 45 participants who received treatment are included in the adverse event reporting.
Arm/Group | APC Flash-Free Adhesive Coated Appliance System | APC II Adhesive Coated Appliance System
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2013-05-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT02030002/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2013-05-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT02030002/Prot_SAP_001.pdf